CLINICAL TRIAL: NCT05780606
Title: Single-cell Transcriptome Identification of UV- and Visible-light-induced Genes in Human Melanocytes in Vivo
Acronym: melatrans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22-PP-22
Record Dates: First submitted 2023-03-10; First posted 2023-03-22 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Skin Diseases
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Voluntary (Other)
  Interventions: Other: Exposed to UV

INTERVENTIONS:
Other: Exposed to UV — Two healthy volunteers will be exposed to UV or visible light in the forearm region. Suction bubbles, and skin biopsies will be performed in test areas, suction bubbles for transcriptome, biopsies for immunohistochemistry

SUMMARY:
Medical condition and pathology studied skin pigmentation. Justification / rationale for the study UV are both the physiological stimulus for skin pigmentation and the main etiological factor in melanoma. Recently, visible (blue) light has also been described to induce skin pigmentation, without any obvious pro-carcinogenic effect. Studies have been carried out to identify genes induced by UV in melanocytes and to understand the mechanisms responsible for photo-induced skin pigmentation. However, the rarity of these cells in the epidermis (3% of cells) has so far been an insurmountable obstacle to achieving this goal. The same is true for visible light, for which the data is even more patchy. The advent of transcriptome analysis techniques at the single cell or single nucleus level will allow us to overcome this obstacle and identify the transcriptional effects of UV and blue light in melanocytes in-situ, as well as in other skin cells (keratinocytes, fibroblasts). Understanding the molecular mechanisms regulated by UV and blue light in melanocytes and other cells will reveal new key steps in skin pigmentation. The data from our study will be used to develop new photoprotective agents as well as new treatments for pigmentary pathologies. Primary objective Describe the variations in gene expression induced by solar ultraviolet (UV) radiation or blue light in human melanocytes in vivo. Secondary objectives Describe the variations in gene expression induced by ultraviolet (UV) radiation sunlight or blue light in other skin cells. Evaluation criteria Single cell transcriptome analysis Immunolabelling on skin sections Population and number of inclusions Healthy male volunteers, phototype III on the Fitzpatrick scale, age 25 + 5 years and of similar corpulence (body mass index between 20 and 28). 2 inclusions Duration of the study Total duration of the study: 12 months Duration of the inclusion phase: 1 month Duration of participation for a patient: 11 days Methodology Two healthy volunteers will be exposed to UV or visible light in the forearm region. Suction blisters, and skin biopsies will be performed in the test areas, suction bubbles for transcriptome, biopsies for immunohistochemistry. The study of gene expression in the different cell types will be done by RNA-Seq on single cells, using the 10X genomics approach. Finally a validation of the results will be carried out by immunostaining with specific antibodies or RNA-Scope. Course of the study - Day 1: The study begins with the determination of the Minimum Erythemal Dose (MED) for each subject in the region of the forearms. This determination will be carried out by means of the administration of six different doses in increasing stages of 25% of UVB + UVA rays (simulated solar ultraviolet spectrum) on six selected test areas (each 1.3 cm²). Exposed areas will be assessed 24 + 2 hours after exposure on Day 2, erythema will be assessed Day 2: Reading of the DEM, and irradiations on two zones in the region of the forearms with respectively a dose of 2 DEM UV, and 48J/cm2 in visible light. A third non-irradiated area will serve as a control. Day 3: A skin blister and biopsy will be performed on each of the three test areas. Cells collected in the blister fluid will be used for the transcriptome and biopsies for validation by immunohistochemistry. Day 11: The subjects will be seen again eight days after the day of sampling, i.e. on Day 11 for removal of sutures and monitoring of healing. On the same day, an evaluation of the level of UV pigmentation induced on each test area will be carried out visually and by colorimetry.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of male sex, phototype III (on the Fitzpatrick scale from I to VI), age 25+5 years and of similar build (body mass index between 20 and 28). - Subject not having been exposed to natural or artificial sunlight in the regions studied for at least 3 months, and not presenting a tan at this level. - Subject showing no skin pathology, scar, or tattoo, in the regions studied. - Subjects who agreed to have a blood test with HIV, hepatitis B and C testing. - Subjects affiliated to a social security scheme - Subjects informed of the aims and nature of the test and having signed a written consent before the start of the study. - Subjects having undergone a general clinical examination attesting to their ability to participate in the study.

Exclusion Criteria:

* - Subjects with a history of dystrophic scarring, particularly of keloids. The preliminary medical examination will endeavor to examine the possible scars of the subject. - Subjects with a dermatological condition that may interfere with assessments. - Subjects with a history of skin cancer. - Subjects having had recourse during the fifteen days preceding the test to systemic or local therapies that risk interfering with the results of the study (eg: corticosteroids, anti-histamines, non-steroidal anti-inflammatory drugs). - Subjects with positive HIV, Hepatitis B (HBSAg surface antigen) and Hepatitis C antibody tests, therefore accepting a blood sample for HIV, hepatitis B and C testing. - Subjects with a history of illness likely, according to the investigator, to put them at risk as a result of the study, in particular photodermatosis, photoaggravated pathologies, atopic dermatitis, chronic urticaria, actinic keratoses, etc. - Subjects allergic to xylocaine adrenaline - Subjects who regularly use sedatives, tranquilizers or other medications known to be photosensitizers - Subjects who have already participated in a pharmacological

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2024-06-13 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Gene expression | 24 hours
  Describe the variations in gene expression induced by solar ultraviolet (UV) radiation or blue light in human melanocytes in vivo

CONTACTS AND LOCATIONS:
Overall Officials: Bahadoran Philippe, PhD, Principal Investigator — CHU de Nice, Service de Dermatologie
Locations (1):
- CHU de Nice - Hôpital de l'Archet, Nice, Alpes-maritimes, France

IPD SHARING:
Plan to Share IPD: No